CLINICAL TRIAL: NCT01694277
Title: A Prospective, Multicenter, Randomized, Open-label, Active-controlled, Two-parallel Groups, Phase 3 Study to Compare the Efficacy and Safety of Masitinib to Sunitinib in Patients With Gastrointestinal Stromal Tumor After Progression With Imatinib at 400mg as First Line Treatment
Brief Title: Masitinib in Patients With Gastrointestinal Stromal Tumour After Progression With Imatinib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AB11002
Record Dates: First submitted 2012-08-22; First posted 2012-09-27 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumour; GIST; non-resectable; metastatic; second line treatment; resistance to imatinib; tyrosine kinase inhibitor
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasm Metastasis | interventions — masitinib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Masitinib (Experimental): Participants receive masitinib (12 mg/kg/day), given orally twice daily.
  Interventions: Drug: Masitinib
- Sunitinib (Active Comparator): Participants receive sunitinib, given at 50 mg/day for 4 consecutive weeks out of 6 weeks, orally
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Masitinib — 12 mg/kg/day
  Other Names: AB1010
  Arms: Masitinib
Drug: Sunitinib — 50 mg/day
  Other Names: Sutent
  Arms: Sunitinib

SUMMARY:
The objective is to compare the efficacy and safety of masitinib at 12 mg/kg/day to sunitinib at 50 mg/day in the treatment of patients with gastro-intestinal stromal tumor (GIST) after progression with imatinib.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor with potent activity against wild-type c-Kit, the juxta membrane domain of c-Kit, and PDGFR. Masitinib is also thought to promote survival via modulation of immunostimulation-mediated anticancer effects and modulation of the tumor microenvironment. The objective is to compare the efficacy and safety of masitinib at 12 mg/kg/day with respect to sunitinib at 50 mg/day in the treatment of imatinib-resistant gastro-intestinal stromal tumor (GIST).

ELIGIBILITY:
Main inclusion criteria include:

* Patient with histological proven metastatic GIST or non-operable locally advanced GIST
* Patient with c-Kit (CD117) positive tumor detected immuno-histochemically
* Patient after at least one progression with imatinib at a dose up to 800mg. Progression is defined as a RECIST 1.1 and/or CHOI disease progression while receiving imatinib treatment.

Main exclusion criteria include:

* Patient treated for a cancer other than GIST within 5 years before enrolment, with the exception of basal cell carcinoma or cervical cancer in situ
* Patient with active central nervous system (CNS) metastasis or with history of CNS metastasis
* Pregnant, or nursing female patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2012-04; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | From day of randomization to death, assessed for a maximum of 60 months
  Overall survival is defined as time in months from the randomization date to the date of death due to any cause. If a patient is not known to have died, then OS will be censored at the date of last known date patient alive.

SECONDARY OUTCOMES:
Survival rate | Every 12 weeks until study completion, assessed for a maximum of 60 months
  Survival rate is defined as the number of patients alive divided by the number of patients in the population of analysis. Assessed at week-8, -16, -24, and every 12 weeks thereafter.
Progression Free Survival (PFS) | From day of randomization to disease progression or death, assessed for a maximum of 60 months
  Progression Free Survival is defined as the time from the randomization date until the date of earliest evidence of disease progression or death, for participants who progressed or died before subsequent cancer therapy. Disease progression will be assessed by the investigator on CT scan according to RECIST 1.1 criteria and/or CHOI criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Axel Le Cesne, M.D., Ph.D, Principal Investigator — Institute Gustave Roussy
Locations (5):
- Washington University School of Medicine, St Louis, Missouri, United States
- France (2):
  - Institut Bergonié, Bordeaux
  - Hôpital l'Archet 2- Service de Cancérologie Digestive, Nice
- Istituto per la Ricerca e la Cura del Cancro (IRCC), Candiolo, Italy
- Erasmus University Medical Center, Rotterdam, Netherlands